CLINICAL TRIAL: NCT00004997
Title: The Experimental Treatment of Transfusion Dependent 5q Minus Syndrome With Leucovorin
Brief Title: Leucovorin for the Treatment of 5 q Minus Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980101; 98-CC-0101
Record Dates: First submitted 2000-03-22; First posted 2000-03-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-07

CONDITIONS: 5q Minus Syndrome; Myelodysplastic Syndrome
Keywords: Hematopoietic; DHFR Enzyme; Anemia; Folic Acid; MDS; Myelodysplasia; Myelodysplastic
MeSH Terms: conditions — Chromosome 5q Deletion Syndrome; Myelodysplastic Syndromes; Anemia; Anemia, Refractory, with Excess of Blasts | interventions — Leucovorin

INTERVENTIONS:
Drug: Leucovorin

SUMMARY:
The 5 q minus syndrome is a condition that occurs due to a missing segment of chromosome 5 in the normal genetic make-up of the cells responsible for forming blood cells. The condition causes patients to have the inability to make blood normally. Many patients with this syndrome need transfusions of red blood cells, platelets, and/or white blood cells. Low levels of platelets may cause the patient to bleed easily and low levels of whit blood cells make the patient susceptible to infections. A small number of patients with 5 q minus syndrome develop leukemia, which is often untreatable with chemotherapy.

Researchers believe that one of the genes missing in 5 q minus syndrome is the gene responsible for making folic acid active in the body. Folic acid is a vitamin required for normal blood production.

The purpose of this study to test the effectiveness of a drug called leucovorin for the treatment of 5 q minus syndrome. Leucovorin is an active form of the vitamin folic acid that does not require the missing genes to activate it.

Patients participating in this study may or may not improve with leucovorin treatment. However, the study will improve researchers understanding of the disease and may lead other potential therapies for the disease.

DETAILED DESCRIPTION:
The objective of this protocol is to determine whether leucovorin treatment can normalize hematopoietic cell growth and differentiation in patients with 5q- syndrome which may lack the gene for dihydrofolate reductase enzyme.

ELIGIBILITY:
All patients 18 years old and older with RA, RARS and RAEB who have a 5q deletion as their sole cytogenetic abnormality who require transfusion support with blood defined as needing at least one unit of packed red blood cells per month for greater than or equal to 2 months and/or thrombocytopenia defined as a platelet count less than 50,000, and/or severe neutropenia (absolute neutrophil count less than 500) are eligible, including patients that had been treated with chemotherapy or experimental agents such as retinoids, phenylbutyrate, amifostine, Vitamin D, ATG or hematopoietic growth factors.

Patients must not be transforming to acute leukemia (greater than 20% blasts in marrow aspirate).

Patients must not have had treatment with growth factors or any other experimental drug within 4 weeks prior to entry on protocol.

Patients must not have an ECOG performance status greater than 2.

Patients must not have an active uncontrolled infection.

No patients for whom bone marrow transplant is indicated as primary therapy.

Must be able to give informed consent.

Patients must not be HIV positive.

Patients must not be pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14
Dates: Start 1998-04; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Mathew P, Tefferi A, Dewald GW, Goldberg SL, Su J, Hoagland HC, Noel P. The 5q- syndrome: a single-institution study of 43 consecutive patients. Blood. 1993 Feb 15;81(4):1040-5. PMID 8427985
- [Background] Funanage VL, Myoda TT, Moses PA, Cowell HR. Assignment of the human dihydrofolate reductase gene to the q11----q22 region of chromosome 5. Mol Cell Biol. 1984 Oct;4(10):2010-6. doi: 10.1128/mcb.4.10.2010-2016.1984. PMID 6504041
- [Background] Maurer BJ, Carlock L, Wasmuth J, Attardi G. Assignment of human dihydrofolate reductase gene to band q23 of chromosome 5 and of related pseudogene psi HD1 to chromosome 3. Somat Cell Mol Genet. 1985 Jan;11(1):79-85. doi: 10.1007/BF01534737. PMID 3856332